CLINICAL TRIAL: NCT06035224
Title: A Single Arm, Phase II Trial of Cadonilimab (AK104) Plus Lenvatinib in Previous Immunotherapy Treated Advanced/Metastatic Clear Cell Renal Cell Carcinoma (ccRCC)
Brief Title: A Study of Cadonilimab（AK104） Plus Lenvatinib in Previous Immunotherapy Treated Advanced/Metastatic Clear Cell Renal Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: Ruijin Hospital (Other); Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLEAR-IT
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Clear Cell Renal Cell Carcinoma、Resistance to Immunotherapy
Keywords: AK104; Lenvatinib

STUDY DESIGN:
Intervention Model Description: A Single Arm, Phase II Trial of Cadonilimab (AK104) Plus lenvatinib in Previous immunotherapy treated Advanced/Metastatic Clear Cell Renal Cell Carcinoma (ccRCC)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK104 combine with lenvatinib (Experimental): Patients will receive AK104 (10mg/kg ,Q3W，intravenously) plus lenvatinib(<60kg，8 mg qd；≥60kg，12mg qd, orally.
  Interventions: Drug: AK104（anti-PD-1/CTLA-4 bi-specific antibody ，intravenously）,lenvatinib（ targeted VEGFR 1-3、FGFR、PDGFRα， small molecule TKI，orally

INTERVENTIONS:
Drug: AK104（anti-PD-1/CTLA-4 bi-specific antibody ，intravenously）,lenvatinib（ targeted VEGFR 1-3、FGFR、PDGFRα， small molecule TKI，orally — AK104 (10mg/kg ,Q3W，intravenously) plus lenvatinib(<60kg，8 mg qd；≥60kg，12mg qd, orally.

SUMMARY:
This is a Phase II, open-label, single arm trial to evaluate the efficacy and safety of AK104 in combination with lenvatinib in previous immunotherapy treated advanced/metastatic clear cell renal cell carcinoma (ccRCC). Subjects with unresectable advanced clear cell renal cell carcinoma (ccRCC) who were second line patients after first-line immunotherapy combined treatment progression. Subjects will receive Cadonilimab（AK104） plus lenvatinib until disease progression, development of unacceptable toxic effects, death, a decision by the physician or patient to withdraw from the trial. The primary endpoint is ORR per RECIST v1.1 as assessed by investigators.

DETAILED DESCRIPTION:
This trial is a single-arm, multicenter clinical study with the aim of enrolling 28 patients with unresectable advanced ccRCC. The study was divided into three research centers, namely Renji Hospital Affiliated to Shanghai Jiao Tong University, Zhongshan Hospital Affiliated to Fudan University in Shanghai, and Shanghai Ruijin Hospital. Lenvatinib capsules are taken orally, 8 mg once daily (qd) for subjects weighing < 60 kg, 12 mg once daily (qd) for subjects weighing ≥ 60 kg, combined with cardunilimab, intravenous infusion, 10 mg/kg, once every three weeks (q3w) until disease progression, death, intolerable toxicity, withdrawal of informed consent, initiation of new antitumor therapy, investigator decision, loss to follow-up, whichever occurs first. Tumor efficacy will be assessed at baseline, every 6 weeks (6 weeks ± 7 days) during treatment, and at end-of-treatment visits.

The experiment is mainly divided into the effectiveness import stage and the cohort expansion stage. The safety introduction phase planned to enroll 12 patients, and after the first dose, the dosing regimen: lenvatinib capsules orally, 8 mg once daily (qd) for subjects weighing < 60 kg, 12 mg once daily (qd) for subjects weighing ≥ 60 kg, in combination with cartunilimab, intravenous infusion, 10 mg/kg every three weeks (q3w), evaluated in 12 patients, 2 or more patients achieved remission before cohort expansion.

The cohort expansion phase plans to enroll 16 patients with accRCC with lenvatinib capsules orally 8 mg once daily (qd) for subjects weighing < 60 kg, 12 mg once daily (qd) for subjects weighing ≥ 60 kg, plus cardunilimab, intravenous infusion, 10 mg/kg every three weeks (q3w) until disease progression, intolerable toxicity, withdrawal of informed consent, loss to follow-up or death, The investigator or subject decided to terminate the treatment, or the study ended the capsules used in this study were donated by Jiangsu Simcere Zaiming Pharmaceutical Co., Ltd., and cardunilimab was donated by Akeso.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent/assent for the trial.
2. Be ≥18 and ≤ 75 years of age on day of signing informed consent. 3）Have histologically or cytologically confirmed diagnosis of RCC with advanced/metastatic disease with clear cell component.

4)Have previous immunotherapy combined treatment progression（ only second line systemic therapy for advanced RCC included) 5)Have measurable disease per RECIST 1.1 as assessed by the investigator /site radiologist.

6)Have estimated life expectancy of at least 3 months. 7)Have ECOG PS 0-1. 8)Hematology: i. absolute neutrophil count (ANC) ≥ 1.5 × 109/L ; ii. platelets ≥ 100 × 109/L ; iii. hemoglobin ≥ 90 g/L.

9)Renal: i. calculated creatinine clearance * (CrCl) ≥ 60 mL/min; * CrCl will be calculated using the Cockcroft-Gault formula CrCL (mL/min) = {(140-age) × body weight (kg) × F }/(SCr (mg/dL) × 72) ii. urine protein < 2 + or 24-hour urine protein must be < 2.0 g.

10)Hepatic: i. serum total bilirubin (TBil) ≤ 1.5 × ULN; ii. AST and ALT ≤ 3 × ULN, ≤ 5 × ULN with liver metastasis; iii. serum albumin (ALB) ≥ 28 g/L.

11)Coagulation function: i. international normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN.

Exclusion Criteria:

1. Has history of allergies to monoclonal antibodies, any components of cadonilimab and lenvatinib
2. Has a known additional malignancy that has progressed or has required active treatment. Note: Subjects with basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or carcinoma in situ are not excluded.
3. Has prior Dual immunotherapy treatment (any anti-PD-1/PD-L1 combined with anti-CLTA-4 ).
4. Has Uncontrolled clinical symptoms or diseases of the heart
5. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 14 days （prednisone>10 mg/day or equivalent dose)
6. Has active autoimmune disease that might deteriorate when receiving an immunostimulatory agents. Subjects with diabetes type I, vitiligo, psoriasis, hypo-or hyperthyroid disease not requiring immunosuppressive treatment are eligible.
7. Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
8. Has an active tuberculosis and syphilitic infection.
9. Has a known history of Human Immunodeficiency Virus (HIV) infection (HIV antibodies).
10. Has known active Hepatitis B (e.g., Hepatitis B surface antigen [HBsAg] reactive and HBV-DNA>500 IU/ml) or Hepatitis C virus (e.g., HCV RNA [qualitative] is detected).
11. Has never recovered from previous anti-tumor treatment toxicity
12. Has active bleeding disorder or other history of significant bleeding episodes .
13. drug abuse and medical, psychological or social conditions that may interfere with patients' participation in research or affect the evaluation of results;
14. Is pregnant or breastfeeding, or expecting to conceive children duration of the trial.

    -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-08-23 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
ORR per RECIST v1.1 as assessed by investigators | Up to 2 years
  ORR is the proportion of subjects with complete response(CR) or partial response(PR) , based on RECIST v1.1

SECONDARY OUTCOMES:
Duration of response (DOR) | Up to 2 years
  Duration of response (DOR) assessed according to RECIST v1.1
Disease control rate (DCR) | Up to 2 years
  Disease control rate (DCR) assessed according to RECIST v1.1
Time to response（TTR） | Up to 2 years
  Time from randomization to obtaining clinical efficacy (CR/PR)
Progression-free survival (PFS) | Up to 2 years
  PFS is defined as the time from the the start of treatment till the first documentation of disease progression (per RECIST v1.1 criteria) assessed by the investigator or death due to any cause (whichever occurs first).
Overall survival (OS) | Up to 2 years
  Overall survival is defined as the time from the start of treatment until death due to any cause.

OTHER OUTCOMES:
Adverse Event | Up to 2 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0, also types and degree
HRQoL based on EORTC QLQ-C30 | Up to 2 years
HRQoL based on EORTC QLQ-H&N35. | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No